CLINICAL TRIAL: NCT05936320
Title: A Randomised Controlled Trial Evaluating Hearing Aid Knowledge and the Effects of Information Leaflets With and Without Illustrations
Brief Title: Evaluating the Effects of Information Leaflets in Adult Aural Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horselvarden Region Ostergotland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bildstöd
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Hearing Impairment
Keywords: aural rehabilitation; hearing aid functions; hearing aid knowledge; information leaflet; visual aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Verbal information along with information leaflets containing text with illustrations about hearing aid functions
  Interventions: Behavioral: Information leaflets with illustrations about hearing aid functions
- Control group (Experimental): Verbal information along with information leaflets containing text-only about hearing aid functions
  Interventions: Behavioral: Information leaflets with only text about hearing aid functions

INTERVENTIONS:
Behavioral: Information leaflets with illustrations about hearing aid functions — The information leaflet contains written information with simple illustrations about placement in noisy environments, how to use a telecoil and about directional microphones function in hearing aids. The time spent presenting the information leaflet was approximately ten minutes.
  Arms: Intervention group
Behavioral: Information leaflets with only text about hearing aid functions — The information leaflet contains written information about placement in noisy environments, how to use a telecoil and about directional microphones function in hearing aids. The time spent presenting the information leaflet was approximately ten minutes.
  Arms: Control group

SUMMARY:
Knowledge about how to manage hearing aids is an important factor in hearing aid success, but studies show that this knowledge ranges from good to poor, even among experienced adult hearing aid users. Information leaflets is a common tool in healthcare to give information with the purpose to increase theoretical knowledge and change behaviour, and illustrations in these leaflets can provide additional understanding for all kinds of patients.

The primary aim of this aural rehabiliation study was to evaluate participants' knowledge about placement in a noisy environment, directional microphone and telecoil function at baseline and postintervention and assessing their perceptions of the benefits of an information leaflet. Additional aim was to investigate whether, an information leaflet with illustrations and accompanying text about hearing aid functions have additional effects on participants' knowledge compared to an information leaflet without illustrations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 years old) with hearing aids from 2012 or later

Exclusion Criteria:

* Hearing aids without possibility to have activated directional microphones and telecoil
* non-swedish speaking (e.g. need interpreter)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Knowledge about hearing aid functions | Baseline, 3 weeks postintervention
  Assessing change in knowledge about placement in noisy environments, telecoil function and directional microphones.
  Open-ended questions where the knowledge assessed by two authors independently of each other, to make the answers quantitative. Interrater reliability was analysed with Cohen's kappa
Perceived benefit | 3 weeks postintervention
  Assessing the perceived benefit of the information leaflet through three items formulated as statements and ranged from (0) not agree at all to (10) completely agree.
  The statements were as follows: 1) the written information I received has increased my understanding of the functions of the hearing aid, and 2) the written information I received has made me better understand how to position myself in different sound environments. If applicable, 3) the written information I received made it easier for me to explain the functions of my hearing aid to a communication partner.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Öberg, Principal Investigator — Horselvarden Region Ostergotland
Locations (1):
- Hearing Clinic of the University Hospital Region Ostergotland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No